CLINICAL TRIAL: NCT00876525
Title: Clinical Investigation of the Freedom SOLO Stentless Heart Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V10604
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Heart Valve Diseases
Keywords: Heart diseases.; Aortic valve diseases.; Aortic valve insufficiency.; Aortic valve stenosis.
MeSH Terms: conditions — Heart Valve Diseases; Heart Diseases; Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, multicenter trial
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Freedom SOLO stentless valve (Other): Prospective data collection on the outcomes in patients treated with the CE Marked Freedom Solo Valve within the approved indication.
  Interventions: Device: Surgical Replacement of the diseased native aortic heart valve with the Freedom SOLO Valve prosthesis

INTERVENTIONS:
Device: Surgical Replacement of the diseased native aortic heart valve with the Freedom SOLO Valve prosthesis — The Freedom SOLO prosthesis is designed for implantation in a supra-annular, sub-coronary position, with a single suture line.

SUMMARY:
This is a trial to demonstrate the safety and effectiveness of the Freedom SOLO heart valve when used to replace a diseased or dysfunctional aortic valve or aortic valve prosthesis.

DETAILED DESCRIPTION:
Freedom SOLO study is a prospective, non-randomized, multicenter trial on the Freedom SOLOvalve implanted in patients requiring aortic valve replacement. The study was conducted at 18 centers in Europe.

The study was based on single sample hypothesis testing that allows comparison of observed morbid event rates to objective performance criteria (OPCs). Based on the guidelines established by the U.S. Food and Drug Administration (FDA), the minimum sample size for this study was 800 valve-years, which is the minimum amount of data needed to test against the OPC of 1.2 %/patient-year.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female 18 years old or older.
* The patient is willing to sign the informed consent.
* The patient which preoperative evaluation indicated the need for native or prosthetic aortic valve replacement.
* Any patient amenable to aortic valve replacement with biological prosthesis should be enrolled in the study, even in conjunction with valve repair, coronary artery bypass grafting and other procedures.
* The patient is located in a geographic location that will enable the subject to return to the study site for all follow-up examinations (i.e. geographically stable).
* Patient will be available to the investigator(s) for postoperative follow-up beyond one year.

Exclusion Criteria:

* The patient has preexisting valve prosthesis in the mitral, pulmonary or tricuspid position.
* The patient requires a double or triple valve replacement (a valve repair is not considered an exclusion criterion).
* The patient has a previously implanted SOLO valve, within the clinical study, that requires replacement.
* The patient has active endocarditis.
* The patient is or will be participating in a concomitant research study of an investigational product.
* The patient is a minor, intravenous drug user, alcohol abuser, prisoner, institutionalized, or is unable to give informed consent.
* The patient has a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy of less than 1 year, or the implant of the device produces an unacceptable increased risk to the patient.
* The patient is pregnant or lactating.
* Patients with congenital bicuspid aortic valve.
* Patients are known to be noncompliant or are unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The complication and survival rates for the Freedom SOLO stentless valve. | up to 1 year
  Safety of the Freedom SOLO was evaluated based on the following adverse events related to cardiac valve replacement: valve thrombosis, thromboembolism, bleeding, anticoagulant-related bleeding, paravalvular leak, endocarditis, clinically significant hemolysis, nonstructural dysfunction, structural valve deterioration, reoperation, explant, and death.
The complication and survival rates for the Freedom SOLO stentless valve. | up to 5 year
  Safety of the Freedom SOLO was evaluated based on the following adverse events related to cardiac valve replacement: valve thrombosis, thromboembolism, bleeding, anticoagulant-related bleeding, paravalvular leak, endocarditis, clinically significant hemolysis, nonstructural dysfunction, structural valve deterioration, reoperation, explant, and death.

SECONDARY OUTCOMES:
Hemodynamic performance of the Freedom SOLO stentless valve: transvalvular peak and mean pressure gradients | up to 5 year
  Decrease of transvalvular peak and mean pressure gradients from preoperative to follow up
Hemodynamic performance of the Freedom SOLO stentless valve: effective orifice area (EOA) in cm2 by transthoracic echocardiography | up to 5 year
  Increase of effective orifice area (EOA) from preoperative to follow up
Hemodynamic performance of the Freedom SOLO stentless valve: EOA index (EOAI cm2/m2). | up to 5 year
  Increase of effective orifice area index from preoperative to follow up.
Hemodynamic performance of the Freedom SOLO stentless valve: cardiac output (CO) Clinically significant improvement in overall patient condition. | up to 5 year
  Improvement of Cardiac Output
Hemodynamic performance of the Freedom SOLO stentless valve: cardiac index (CI) Clinically significant improvement in overall patient condition. | up to 5 year
  Improvement of Cardiac Index
Hemodynamic performance of the Freedom SOLO stentless valve: regurgitation Clinically significant improvement in overall patient condition. | up to 5 year
  Evaluation of regurgitation, location and severity
Preoperative and postoperative NYHA functional classifications | Preoperatively, after the procedure (1 week), 3-6 months, 12 months and annually thereafter
  NYHA functional classification data is presented as the number and percentage of patients in each functional class.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Thalmann, MD, Principal Investigator — KH Hietzing Wien
Locations (19):
- Austria (2):
  - Krankenhaus Hietzing, Vienna
  - Medical University Vienna, Vienna
- Belgium (2):
  - St. Luc Hospital, Brussels
  - University Hospital Gent, Ghent
- France (2):
  - Hôpital Pontchaillou - CHU, Rennes
  - Hôpital Trousseau - CHRU, Tours
- Germany (4):
  - Herz- und Gefäß-Klinik GmbH, Bad Neustadt an der Saale
  - Charité Hospital, Berlin
  - Herzzentrum Dresden Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Erlangen, Klinik für Herzchirurgie, Erlangen
- Italy (3):
  - Ospedale del Cuore, Fondazione G. Monasterio, Massa
  - Ospedale "S. Maria di Ca' Foncello", Treviso
  - Ospedale S. Maria Della Misericordia, Udine
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Thoraxcentrum, Enschede
  - University Hospital St. Radboud, Nijmegen
- Hospital S. João, Porto, Portugal
- Inselspital, University Hospital Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thalmann M, Grubitzsch H, Matschke K, Glauber M, Tan E, Francois K, Amorim MJ, Hensens AG, Cesari F, Feyrer R, Diegeler A, Veit F, Repossini A; Freedom Solo Investigators. A European Multicenter Study of 616 Patients Receiving the Freedom Solo Stentless Bioprosthesis. Ann Thorac Surg. 2016 Jan;101(1):100-8. doi: 10.1016/j.athoracsur.2015.06.096. Epub 2015 Oct 9. PMID 26443880